CLINICAL TRIAL: NCT00997048
Title: Comparison Between Laying Open and Sinus Excision of Pilonidal Sinus - a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Professor Wilhelm Graf, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPN 2002/139
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laying open (Experimental)
  Interventions: Procedure: Laying open
- Sinus excision (Active Comparator)
  Interventions: Procedure: Sinus excision

INTERVENTIONS:
Procedure: Laying open — Laying open Antibiotics Dalacin 300 mg tablets or iv infusion 600 mg
  Arms: Laying open
Procedure: Sinus excision — Sinus excision Antibiotics Dalacin tablets 300 mg or iv infusion 600 mg
  Arms: Sinus excision

SUMMARY:
A pilonidal sinus is a cyst or abscess near or on the natal cleft of the buttocks that often contains hair and skin debris. The condition is common and requires surgery to be cured. Several surgical procedures are described in literature. The most common surgical procedure in Sweden is excision of the sinus followed by suturing the subcutaneous tissue and skin. This method, however, has some problems regarding healing and recidives. Therefore this study is comparing the standard excision procedure to another surgical procedure, laying open. Healing frequency is the main variable, but postoperative pain, sick leave time and patient satisfaction is also measured.

ELIGIBILITY:
Inclusion Criteria:

* Pilonidal sinus eligible for surgery
* Age > 18 years
* Swedish speaking

Exclusion Criteria:

* Active signs of infection prohibiting primary sewing of the wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Healing frequency | 12 months

SECONDARY OUTCOMES:
pain according to a visual analogue scale | 7 days
scar/wound length | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Graf, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, surgery, Uppsala, Sweden

REFERENCES:
- [Derived] Lorant T, Ribbe I, Mahteme H, Gustafsson UM, Graf W. Sinus excision and primary closure versus laying open in pilonidal disease: a prospective randomized trial. Dis Colon Rectum. 2011 Mar;54(3):300-5. doi: 10.1007/DCR.0b013e31820246bf. PMID 21304300